CLINICAL TRIAL: NCT04767737
Title: The Effect of Topically Administered Lavender Aromatherapy on the Pain of Insulin Injection in Diabetic Patients: A Double-Blind Randomized Controlled Clinical Trial
Brief Title: The Effect of Aromatherapy on the Insulin Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Hatice Demirağ, Principal Investigator, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RCT1004201704062014
Record Dates: First submitted 2020-11-26; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Pain; Aromatherapy; Subcutaneous Injections
Keywords: Pain; aromatherapy; topical lavender oil; subcutaneous injections
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The sample was determined as 159 (53 for each group) patients for three groups (lavender oil group, placebo group, control group) by using the power analysis method (G*Power 3.1.9.6 program), with the margin of error α=0.05, 0.25 medium effect size, and 0.80 (80%) target strength of the test. However, 7 patients who met the study inclusion criteria were added to each group (60 in the lavender oil group, 60 in the placebo group, 60 in the control group) in case some of the participants quit the study for any reason (Figure 1). While the patients were randomized, different application groups (topical lavender oil, placebo, control group) were determined by lot in different months (May, June, and July) to minimize the possibility of being affected by each other.
Who Masked: Participant, Care Provider
Masking Description: Since this study was a double-blind randomized controlled study, no information about the drug (topical lavender oil, topical water) was given to the nurse (researcher) who gave insulin injection, and the patient to reduce bias. The drug to be used was applied in spray bottles without any labels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical lavender oil group (Experimental): Before the administration, pain level, blood pressure, respiratory rate, pulse rate, oxygen saturation level (SPO2), and blood glucose of all patients (topical lavender oil, placebo, and control groups) were measured, and then, 3 puffs (0.3 ml) of 100% lavender (Lavandula Angustifolia) essential oil to the topical lavender oil group were sprayed on the arms of the patients. 5 minutes later, the insulin injection site was wiped with 10% povidone-iodine (baticonol) in all patients, and the injection was given. During the administration of the insülin, the pain levels of the patients were measured again. After giving the injection, blood pressure, respiratory rate, pulse rate, oxygen saturation level, and blood glucose of the patients were also measured again.
  Interventions: Other: Topically Administered Lavender Aromatherapy
- Placebo group (Placebo Comparator): Before the administration, pain level, blood pressure, respiratory rate, pulse rate, oxygen saturation level (SPO2), and blood glucose of all patients (topical lavender oil, placebo, and control groups) were measured, and then, 3 puffs (0.3 ml) of topical distilled water to the placebo group were sprayed on the arms of the patients. No application was applied to the control group. 5 minutes later, the insulin injection site was wiped with 10% povidone-iodine (baticonol) in all patients, and the injection was given. During the administration of the insülin, the pain levels of the patients were measured again. After giving the injection, blood pressure, respiratory rate, pulse rate, oxygen saturation level, and blood glucose of the patients were also measured again.
  Interventions: Other: Topically Administered Water
- Control groups (No Intervention): Before the administration, pain level, blood pressure, respiratory rate, pulse rate, oxygen saturation level (SPO2), and blood glucose of all patients (topical lavender oil, placebo, and control groups) were measured.No application was applied to the control group. 5 minutes later, the insulin injection site was wiped with 10% povidone-iodine (baticonol) in all patients, and the injection was given. During the administration of the insülin, the pain levels of the patients were measured again. After giving the injection, blood pressure, respiratory rate, pulse rate, oxygen saturation level, and blood glucose of the patients were also measured again.

INTERVENTIONS:
Other: Topically Administered Lavender Aromatherapy — 3 puffs (0.3 ml) of 100% lavender (Lavandula Angustifolia) essential oil to the topical lavender oil group were sprayed on the arms of the patients.
  Arms: Topical lavender oil group
Other: Topically Administered Water — 3 puffs (0.3 ml) of topical distilled water to the placebo group were sprayed on the arms of the patients.
  Arms: Placebo group

SUMMARY:
Needle phobia occurs in more than half of diabetic patients due to the pain caused by frequent insulin injection. Therefore, this study evaluated the effect of topically administered lavender aromatherapy on the pain of insulin injection in diabetic patients.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a serious chronic disease that negatively affects the quality of life. To control the course of the disease and to reduce its complications, insulin treatment is planned for the whole life of Type 1 diabetic patients, and frequently for approximately 40% of Type 2 diabetic patients. Frequent or incorrect administration of insulin injections may lead to the development of complications such as regional pain, ecchymosis, or hematoma on the injection site. It is emphasized that the pain caused by repeated insulin injections negatively affects the psychological well-being of the individuals as well as their physical comfort. Pain control is one of the main tasks of nurses. By alleviating pain, the patient's acceptance of treatment increases, and thus the quality of life improves. In the literature, lavender is reported to have the ability to heal burns and insect bites as well as analgesic, wound healing, antibacterial, antifungal, sedative, and antidepressant effects. The main components of lavender, such as lavender and linalyl acetate and linalool, are also recommended as topical analgesics in animal models. Whatever the cause, acute pain is a serious problem for individuals with chronic illnesses. Therefore, this study evaluated the effect of topically administered lavender aromatherapy on the pain of insulin injection in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years of age or older,
* having Type-1 DM or Type-2 DM disease,
* being conscious and communicating, not having mental and cognitive impairment,
* not having eczema and fragrance allergy to lavender,
* not having an alcohol or narcotic addiction,
* not having a head injury or convulsion history,
* not having a diabetes-related neuropathy, and
* if the patient took sedatives or analgesics, at least 6 hours would pass,

Exclusion Criteria:

* having a history of addiction or diagnosed psychological disorders,
* having an unstable hemodynamic status,
* having skin disease symptoms such as wounds and eczema at the insulin injection site and,
* having an allergy to lavender.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Pain Level before insulin injection | day 1
  It was evaluated between the Verbal Category Scale (VCS) pain scores of the patients in the topical lavender oil group before insulin injection. Verbal Category Scale is based on the patient's choice of the most appropriate word to identify his/her pain. Accordingly, the patient was asked to rate his/her pain between 0-4 as 0; no pain, 1: mild pain, 2: severe pain, 3: very severe pain, 4: unbearable pain.
Pain Level before insulin injection | day 1
  It was evaluated between the Visual Analogue Scale (VAS) pain scores of the patients in the topical lavender oil group before insulin injection. Visual Analogue Scale is used to digitalize the pain level that cannot be measured numerically. A line with a length of 100 mm has the words "no pain" at one end and "the most unbearable pain" on the other. The patient indicates his/her pain by choosing the most appropriate place on the line. Then, the level of pain experienced by the patient is determined by using a scale with scores between 0-10. According to this scoring system, less than 3 points indicate mild pain, 3-6 points indicate moderate pain, and more than 6 points indicate severe pain.
Pain Level after insulin injection | day 1
  It was evaluated between the VCS pain scores of the patients in the topical lavender oil group during insulin injection. Verbal Category Scale is based on the patient's choice of the most appropriate word to identify his/her pain. Accordingly, the patient was asked to rate his/her pain between 0-4 as 0; no pain, 1: mild pain, 2: severe pain, 3: very severe pain, 4: unbearable pain.
Pain Level after insulin injection | day 1
  It was evaluated between the VAS pain scores of the patients in the topical lavender oil group during insulin injection. Visual Analogue Scale is used to digitalize the pain level that cannot be measured numerically. A line with a length of 100 mm has the words "no pain" at one end and "the most unbearable pain" on the other. The patient indicates his/her pain by choosing the most appropriate place on the line. Then, the level of pain experienced by the patient is determined by using a scale with scores between 0-10. According to this scoring system, less than 3 points indicate mild pain, 3-6 points indicate moderate pain, and more than 6 points indicate severe pain.
Blood glucose before insulin injection | day 1
  Before the administration blood glucose (mg/dl) of all patients (topical lavender oil, placebo, and control groups) were measured. Blood glucose measurement is done with a blood glucose meter (glucometer) and a measuring stick (strip). Fasting blood glucose 70-125 mg / dl was considered normal.
Oxygen Saturation (SPO2) before insulin injection | day 1
  Before the administration oxygen saturation level (SPO2)(%) of all patients (topical lavender oil, placebo, and control groups) were measured. The researcher measured the oxygen saturation in subcutaneous arterial blood with a "Pulse oximeter" device that is reliable, easy to use, does not require calibration and does not cause pain to the patient in its application. Normal value of oxygen saturation (SpO2) (%) was accepted as 96-98%. After placing a probe in the periphery (on the patient's finger) by the investigator, the signal received from the periphery and the value on the image screen (monitor) where the pulse wave sample was projected was recorded as oxygen saturation.
Systolic and Diastolic Blood Pressure before insulin injection | day 1
  Before the administration blood pressure (mm/Hg) of all patients (topical lavender oil, placebo, and control groups) were measured. Blood Pressure Measurement was performed using a conventional cuffed sphygmomanometer that can measure systolic and diastolic blood pressure, whose reliability was approved according to international standards and calibrated by the company in technical laboratories for certain periods. The cuff of the sphygmomanometer will be inflated to 20 mm / Hg above the systolic pressure by tying it to cover 2/3 of the arm, and the measurement will be carried out by the researcher.
Pulse rate before insulin injection | day 1
  Before the administration pulse rate (min) of all patients (topical lavender oil, placebo, and control groups) were measured. The pulse was obtained by the investigator palpating the superficial arteries (by touching them with the hand) and counting the beats felt for one minute. 60 to 100 beats per minute was considered normal for an adult.
Respiration rate before insulin injection | day 1
  Before the administration Respiration rate (min) of all patients (topical lavender oil, placebo, and control groups) were measured. Respiration rate was measured by the number of diaphragm movements per minute. For an adult at rest, 12 to 20 per minute was considered normal for respiratory rate.
Blood glucose after insulin injection | day 1
  After the administration blood glucose (mg/dl) of all patients (topical lavender oil, placebo, and control groups) were measured. Blood glucose measurement is done with a blood glucose meter (glucometer) and a measuring stick (strip). Fasting blood glucose 140-199 mg / dl was considered normal.
Oxygen Saturation (SPO2) after insulin injection | day 1
  After the administration oxygen saturation level (SPO2)(%) of all patients (topical lavender oil, placebo, and control groups) were measured. The researcher measured the oxygen saturation in subcutaneous arterial blood with a "Pulse oximeter" device that is reliable, easy to use, does not require calibration and does not cause pain to the patient in its application. Normal value of oxygen saturation (SpO2) (%) was accepted as 96-98%. After placing a probe in the periphery (on the patient's finger) by the investigator, the signal received from the periphery and the value on the image screen (monitor) where the pulse wave sample was projected was recorded as oxygen saturation.
Systolic and Diastolic Blood Pressure after insulin injection | day 1
  After the administration blood pressure (mm/Hg) of all patients (topical lavender oil, placebo, and control groups) were measured. Blood Pressure Measurement was performed using a conventional cuffed sphygmomanometer that can measure systolic and diastolic blood pressure, whose reliability was approved according to international standards and calibrated by the company in technical laboratories for certain periods. The cuff of the sphygmomanometer will be inflated to 20 mm / Hg above the systolic pressure by tying it to cover 2/3 of the arm, and the measurement will be carried out by the researcher.
Pulse rate after insulin injection | day 1
  After the administration pulse rate (min) of all patients (topical lavender oil, placebo, and control groups) were measured. The pulse was obtained by the investigator palpating the superficial arteries (by touching them with the hand) and counting the beats felt for one minute. 60 to 100 beats per minute was considered normal for an adult.
Respiration rate after insulin injection | day 1
  After the administration Respiration rate (min) of all patients (topical lavender oil, placebo, and control groups) were measured. Respiration rate was measured by the number of diaphragm movements per minute. For an adult at rest, 12 to 20 per minute was considered normal for respiratory rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Tecnical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I'll decide later

REFERENCES:
- [Derived] Demirag H, Hintistan S, Bulut E. The effect of topically administered lavender aromatherapy on the pain of insulin injection in diabetic patients: a double-blind randomized controlled clinical trial. Turk J Med Sci. 2022 Dec;52(6):1845-1853. doi: 10.55730/1300-0144.5531. Epub 2022 Dec 21. PMID 36945997